CLINICAL TRIAL: NCT02661607
Title: A Prospective Study to Compare Point of Care Echocardiography Versus Chest Radiography for the Assessment of Central Venous Catheter Placement in Critical Care Environments
Brief Title: Point of Care Echocardiography Versus Chest Radiography for the Assessment of Central Venous Catheter Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Peter Korsten, Dr. med., University of Göttingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1/3/14
Record Dates: First submitted 2015-06-17; First posted 2016-01-22 (Estimated); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Central Venous Catheterization; Ultrasound; Emergency Medicine; Critical Care
MeSH Terms: interventions — Central Venous Catheters; X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Point of care echocardiography after central venous catheter (Other): Point of care echocardiography plus chest radiography
  Interventions: Procedure: Point of care echocardiography; Device: Central venous catheter placement; Procedure: Chest radiography

INTERVENTIONS:
Procedure: Point of care echocardiography — Point of echocardiography is performed after routine placement of central venous catheterization and compared with routine chest radiography
Device: Central venous catheter placement — Central venous catheter placement is performed as per local guidelines in critically ill patients
Procedure: Chest radiography — Routine chest radiography is performed after central venous catheter placement in critically ill patients

SUMMARY:
A prospective study to compare the use of point of care echocardiography versus routine chest radiography for the assessment of central venous catheter placement.

ELIGIBILITY:
Inclusion Criteria:

* patients who require central venous catheterization in critical care environments (ICU, IMC)
* patients (or legal guardian) who provide written informed consents
* patients aged 18 years or older

Exclusion Criteria:

* patients who are unable/unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-10; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Adequate placement of the central venous catheter | 2 hours
  Participants will be followed for the period after the intervention to assess correct placement, an expected average of 2 hours

SECONDARY OUTCOMES:
Time needed for the intervention (bedside echocardiography) | 5 Minutes
  Time of the procedure will be measured, an expected average of 5 minutes
Performance of residents as assessed by the time needed to perform the echocardiography | 5 Minutes
  Time needed to perform the echocardiography will be measured with an expected average of 5 minutes
Time needed for chest radiography to be performed | 2 hours
  Time will be measured after requesting chest radiography via telephone until chest radiographs are available for review, an expected average of 2 hours
Adverse Events | 24 hours
  Patients will be followed as per local guidelines to detect complications by central venous catheter placement, usual time Frame of 24 hours (e. g. pneumothorax from cvc placement)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Korsten, MD, Principal Investigator — University Medical Center Göttingen, Department of Nephrology and Rheumatology
Locations (1):
- University of Göttingen, Göttingen, Germany

REFERENCES:
- [Derived] Korsten P, Mavropoulou E, Wienbeck S, Ellenberger D, Patschan D, Zeisberg M, Vasko R, Tampe B, Muller GA. The "rapid atrial swirl sign" for assessing central venous catheters: Performance by medical residents after limited training. PLoS One. 2018 Jul 16;13(7):e0199345. doi: 10.1371/journal.pone.0199345. eCollection 2018. PMID 30011285